CLINICAL TRIAL: NCT01073059
Title: Open-label, Two-period, One Sequence, Multiple Dose, Crossover Study, A Study to Investigate Pharmacokinetic Interactions in Combination Treatment of Valproic Acid and Ertapenem in Normal Healthy Male Subjects
Brief Title: Pharmacokinetic Interactions in Combination Treatment of Valproic Acid and Ertapenem in Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chonbuk National University (Other)
Responsible Party: Study Director, Chang-Seop Lee, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CUH_2009_VPA
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: valproic acid; ertapenem
MeSH Terms: interventions — Valproic Acid; Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valproic acid (Experimental)
  Interventions: Drug: Valproic acid and Ertapenem

INTERVENTIONS:
Drug: Valproic acid and Ertapenem

SUMMARY:
* This trial is conducted to assess pharmacokinetic characteristics of valproic acid when valproic acid single treatment and valproic acid & ertapenem combination treatment
* This trial is performed to evaluate safety of the combination treatment compare with single treatment
* The investigators carry this trial out to study mechanism of combination treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are healthy volunteers, men 19~50 years
* Subjects who have a weight more then 50kg and a condition ± 20% range of ideal weight

Exclusion Criteria:

* Subjects with evidence of clinically significant hepatic, pancreatic, renal, neurological, pulmonary, endocrine, blood tumor, psychiatric or cardiovascular disease
* Subjects who have a GI disease (crohn's disease, etc.) that would increase the influence with absorbance medication or a GI surgery excluding appendectomy and hernia surgery
* Subjects with uncontrolled hypotension (indicated by a sitting systolic blood pressure≤ 100 mmHg or diastolic blood pressure≤ 65 mmHg measured) and hypertension (indicated by a sitting systolic blood pressure≥ 150 mmHg or diastolic blood pressure≥ 95 mmHg measured) at vital sign measurement
* Subjects with known allergy, hypersensitivity (anaphylaxis-type reaction; especially penicillin antibiotics)
* Subjects with a history of drug abuse
* Subjects who received certain medication (include oriental medicine) within the past 3 weeks or certain OTC-drug within 1 week
* Subjects who participated in other clinical investigation within 2months prior to first administration Subjects who did whole blood donation (within 2months) or apheresis (within 1months) prior to first administration
* Subjects who are chronic drinkers

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08

PRIMARY OUTCOMES:
Maximum Plasma Concentration at Steady State (Cmax ss) in Valproic acid single treatment | serial pharmacokinetic plasma concentrations were drawn at 72, 73, 74, 75, 76, 77, 78, 80, and 84 hours according to protocol
Maximum Plasma Concentration at Steady State (Cmax ss) in Valproic acid and Ertapenem combination treatment | serial pharmacokinetic plasma concentrations were drawn at 144, 145, 146, 147, 148, 149, 150, 152, and 156 hours according to protocol
Area Under the Concentration Versus Time Curve in Valproic acid single treatment | serial pharmacokinetic plasma concentrations were drawn at 72, 73, 74, 75, 76, 77, 78, 80, and 84 hours according to protocol
Area Under the Concentration Versus Time Curve in Valproic acid and Ertapenem combination treatment | serial pharmacokinetic plasma concentrations were drawn at 144, 145, 146, 147, 148, 149, 150, 152, and 156 hours according to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Seop Lee, MD/Prof., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea